CLINICAL TRIAL: NCT01095523
Title: Prospective Randomized Trial Evaluating Mandatory Second Look Surgery With HIPEC and CRS vs. Standard of Care in Subjects at High Risk of Developing Colorectal Peritoneal Metastases
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100037; 10-C-0037
Record Dates: First submitted 2010-03-27; First posted 2010-03-30 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-02-09

CONDITIONS: Colorectal Carcinoma; Peritoneal Carcinomatosis
Keywords: Colon Cancer; Rectal Cancer; Peritoneal Perfusion; Metastatic Cancer; Recurrence; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Peritoneal Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Neoplasm Metastasis; Recurrence

INTERVENTIONS:
Procedure: Laparotomy+ HIPEC +/- CRS

SUMMARY:
Background:

* Survival rates for colorectal cancer depend on a number of factors, including the existence of tumors outside the colon and rectum. Patients who had tumors elsewhere in the abdomen (such as in the peritoneum or ovaries) when they were diagnosed, as well as patients who had bleeding or obstruction when they were diagnosed, have a high risk of cancer recurrence even after surgery or other treatment.
* If additional tumors are discovered early and removed while they are still small (often before they can show up on scans), survival rates may improve. In addition, patients who receive a heated chemotherapy solution delivered directly to the abdomen often have better treatment outcomes regardless of whether additional tumors were found. Further research can help determine the usefulness of both of these treatments in improving the outcomes of patients with colorectal cancer.

Objectives:

- To determine whether patients who have had surgery for colorectal cancer have improved outcomes after receiving additional surgery combined with direct chemotherapy, compared with those who receive the current standard of care.

Eligibility:

- Individuals at least 18 years of age who have had surgery for colorectal cancer within the past 14 months, who are considered to be at high risk for cancer recurrence, and whose current imaging scans show no signs of additional tumors.

Design:

* Participants will be divided into two treatment groups: a surgery group and a standard of care group.
* Participants who had surgery less than 11 months ago will be enrolled in a 3-month lead-in phase to receive standard follow-up care, including labs, scans, and physical examinations, before being randomized to a treatment group between 11 and 14 months after surgery. Participants who had surgery between 11 and 14 months ago will be randomized at the time of enrollment.
* Participants in the surgery group will have the following procedures within 2 weeks of randomization:
* Abdominal surgery where surgeons will look for and remove any tumors and take biopsies to check for cancer cells
* Heated chemotherapy, with three chemotherapy drugs administered directly to the abdomen
* In-patient recovery and follow-up visits beginning 3 to 6 weeks after discharge.
* Participants in the standard of care group will have the standard follow-up schedule for high-risk colorectal cancer patients:
* Clinic evaluations every 3 months for 2 years, and then every 6 months for 3 years and yearly thereafter....

DETAILED DESCRIPTION:
BACKGROUND:

* Peritoneal carcinomatosis (PC) from colorectal cancer (CRC) treated with chemotherapy alone results in median survival of 5 to 13 months.

  .-Approximately, 55% of high risk patients (Patients presenting with synchronous PC, ovarian metastases perforated primary, and emergency presentation with bleeding or obstructing lesions) will develop PC.
* Early PC is undetectable by conventional imaging.
* Cytoreductive surgery (CRS) and hyperthermic intraperitoneal chemotherapy (HIPEC) for early PC from CRC resulted in median survival of 48-63 months and 5 year survival of 51 %.
* This study is a prospective randomized trial designed to answer the question whether mandatory second look surgery (MSLS) with CRS and HIPEC will prolong overall survival when compared to the standard of care.

OBJECTIVES:

Primary Objective:

- To compare the overall survival of patients at high risk for developing PC from CRC who undergo M SLS + HIPEC and CRS (if applicable) vs. similar patients who receive standard of care.

Secondary Objectives:

* To determine recurrence-free survival in both arms.
* To investigate selection criteria for patient who might benefit from a strategy of MSLS with CRS + HIPEC.

ELIGIBILITY:

* Patients who have undergone curative resection f or CRC who are at high risk for recurrence
* Patients who shown no evidence of disease at the time of enrollment
* Patients with ECOG less than or equal to 0-2 and suitable candidates for laparotomy, HIPEC and CRS.

DESIGN:

* High risk CRC patients for developing PC who underwent curative surgery and subsequently received standard of care and remained NED for 12 months after primary surgery will be randomized into MSLS/CRS/HIPEC or continuing standard of care.
* HIPEC will be done using Oxaliplatin/5-FU/Leucovorin.
* Up to 100 patients will be enrolled to allow for 35 evaluable patients in each arm; accrual is expected to last 5 years.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Histologically confirmed colorectal adenocarcinoma.
  2. Curative resection (NED at closure) for CRC which was (1) perforated into the peritoneal cavity, (2) associated with minimal PC which was completely excised at the time of initial operation, (3) T4 lesion that required en bloc resection of additional organs, (4) associated with ovarian metastases or (5) emergency presentation with lesions associated with obstruction and/or bleeding.

     Note: Patient who presented at the time of diagnosis with limited extra abdominal metastases may be eligible if the lesions were completely resected and the patient remains NED.
  3. Received at least 3 months of standard of care adjuvant therapy and is disease free by conventional imaging at time of registration and/or randomization.

     Note: The imaging will be reviewed by an experienced radiologist and a surgical attending prior to enrollment.
  4. Greater than or equal to 18 years of age.
  5. Must be able to understand and sign the Informed Consent
  6. Clinical performance status of ECOG less than or equal to 2.
  7. Life expectancy of greater than three months.
  8. Patients of both genders must be willing to practice birth control during and for four months after receiving chemotherapy.
  9. Hematology:
* Absolute neutrophil count greater than 1500/mm(3) without the support of Filgrastim.
* Platelet count greater than 75,000/mm(3).
* Hemoglobin greater than 8.0 g/dl.

  j. Chemistry:
* Serum creatinine less than or equal to 1.5 mg/dl unless the measured creatinine clearance is greater than 60mL/min/1.73m(2).
* Total bilirubin less than or equal to 2 mg/dl, except for patients with diagnosis of Gilbert's disease or hepatic pedicle obstruction then total bilirubin must be less than or equal to 5 mg/dl.

  k. INR less than or equal to 1.8.

  l. Stable serum CEA levels

  m. No history of prior/other malignancies within the 2 years prior to enrollment with the exception of basal cell carcinoma.

EXCLUSION CRITERIA:

1. Women of child-bearing potential who are pregnant or breast feeding because of the potentially dangerous effects of the chemotherapy on the fetus or infant.
2. Active systemic infections, coagulation disorders or other major medical illnesses precluding major surgery.
3. Prior experimental therapy with novel agents
4. Prior HIPEC
5. History of brain metastases
6. Childs B or C cirrhosis or with evidence of severe portal hypertension by history, endoscopy, or radiologic studies or with evidence of moderate to severe ascites.
7. Weight less than 40 kg.
8. History of congestive heart failure and/or an LVEF < 40%

   Note: Patients at increased risk for coronary artery disease or cardiac dysfunction (e.g., > 65yo, diabetes, history of hypertension, elevated LDL, first degree relative with coronary artery disease) will undergo full cardiac evaluation and will not be eligible if they demonstrate significant irreversible ischemia on stress thallium or an ejection fraction < 40%. Patients may be eligible if cardiac status is treated and improves to within eligibility criteria.
9. Significant COPD or other chronic pulmonary restrictive disease with PFT's indicating an FEV1 less than 50% or a DLCO less than 40% predicted for age.

   Note: Patients who have shortness of breath with minimal exertion or who are at risk for pulmonary disease (e.g., chronic smokers) will undergo pulmonary function testing.
10. Discretion of principle investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01-14; Primary Completion 2012-02-09 (Actual); Study Completion 2012-02-09 (Actual)

PRIMARY OUTCOMES:
To compare the overall survival of patients at high risk for developing peritoneal carcinomatosis from colorectal cancer who undergo mandatory second look surgery + HIPEC and CRS (if applicable) vs. similar patients who receive standard of care. | Follow-up will occur every 3 months for two years, every six months for three ye

SECONDARY OUTCOMES:
To determine recurrence-free survival in both arms. To investigate selection criteria for patients who might benefit from a strategy of MSLS with CRS + HIPEC. | Follow-up will occur every 3 months for two years, every six months for three ye

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Chu DZ, Lang NP, Thompson C, Osteen PK, Westbrook KC. Peritoneal carcinomatosis in nongynecologic malignancy. A prospective study of prognostic factors. Cancer. 1989 Jan 15;63(2):364-7. doi: 10.1002/1097-0142(19890115)63:23.0.co;2-v. PMID 2910444
- [Background] Colucci G, Gebbia V, Paoletti G, Giuliani F, Caruso M, Gebbia N, Carteni G, Agostara B, Pezzella G, Manzione L, Borsellino N, Misino A, Romito S, Durini E, Cordio S, Di Seri M, Lopez M, Maiello E, Montemurro S, Cramarossa A, Lorusso V, Di Bisceglie M, Chiarenza M, Valerio MR, Guida T, Leonardi V, Pisconti S, Rosati G, Carrozza F, Nettis G, Valdesi M, Filippelli G, Fortunato S, Mancarella S, Brunetti C; Gruppo Oncologico Dell'Italia Meridionale. Phase III randomized trial of FOLFIRI versus FOLFOX4 in the treatment of advanced colorectal cancer: a multicenter study of the Gruppo Oncologico Dell'Italia Meridionale. J Clin Oncol. 2005 Aug 1;23(22):4866-75. doi: 10.1200/JCO.2005.07.113. Epub 2005 Jun 6. PMID 15939922
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Murray T, Thun MJ. Cancer statistics, 2008. CA Cancer J Clin. 2008 Mar-Apr;58(2):71-96. doi: 10.3322/CA.2007.0010. Epub 2008 Feb 20. PMID 18287387
- [Derived] Savolainen-Kopra C, Haapakoski J, Peltola PA, Ziegler T, Korpela T, Anttila P, Amiryousefi A, Huovinen P, Huvinen M, Noronen H, Riikkala P, Roivainen M, Ruutu P, Teirila J, Vartiainen E, Hovi T. STOPFLU: is it possible to reduce the number of days off in office work by improved hand-hygiene? Trials. 2010 Jun 4;11:69. doi: 10.1186/1745-6215-11-69. PMID 20525328
- [Derived] Ripley RT, Davis JL, Kemp CD, Steinberg SM, Toomey MA, Avital I. Prospective randomized trial evaluating mandatory second look surgery with HIPEC and CRS vs. standard of care in patients at high risk of developing colorectal peritoneal metastases. Trials. 2010 May 25;11:62. doi: 10.1186/1745-6215-11-62. PMID 20500867